CLINICAL TRIAL: NCT06381895
Title: The Efficacy of Radiomics to Predict Tumor Microenvironment Markers and Comprehensive Therapy for Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-467-01; NCT06442839 (obsolete NCT alias)
Record Dates: First submitted 2024-04-15; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Bladder Cancer; Radiomics; Immunotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Sun Yat-sen Memorial Hospital cohort
- 2: Third Affiliated Hospital of Sun Yat-sen University cohort
- 3: Sun Yat-sen University Cancer Center cohort

SUMMARY:
The aim of this study was to develop an radiomic model based on CT images to evaluate markers of the bladder cancer microenvironment, such as TSR,TIL, and IP. Secondly, the association of the radiomic model with clinical outcomes and immunotherapy response was investigated.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age;
2. Performing TURB-t or RC during 2010-2022;
3. The primary lesion was located in the bladder, and the pathological diagnosis was urothelial carcinoma;
4. Complete clinical information, pathological data, preoperative pelvic enhanced CT and follow-up records;

Exclusion Criteria:

1. Patients with distant metastasis;
2. Combined with other malignant tumors or malignant tumor treatment history
3. Malignant tumors of upper urinary tract;
4. Clinical information, pathological data, preoperative pelvic enhanced CT and follow-up records were missing;
5. Other situations in which the researcher considers it inappropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed primary bladder cancers
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Tumour-infiltrating lymphocytes (TIL) | 1 year
  TILs were evaluated using paraffin-embedded tumour tissue samples stained with H&E according to established protocols.

SECONDARY OUTCOMES:
overall survival | 1 year
  We obtain this data through telephone follow-up and evaluate it according to the date of surgery
cancer-specific survival | 1 year
  We obtain this data through telephone follow-up and evaluate it according to the date of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Liushan Ou, Study Chair — Medical Ethics Committee, Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen K, Li X, Liu L, Wang B, Liang W, Chen J, Gao M, Huang X, Liu B, Sun X, Yang T, Zhao X, He W, Luo Y, Huang J, Lin T, Zhong W. Correlation of noninvasive imaging of tumour-infiltrating lymphocytes with survival and BCG immunotherapy response in patients with bladder cancer: a multicentre cohort study. Int J Surg. 2025 Jan 1;111(1):920-931. doi: 10.1097/JS9.0000000000001999. PMID 40053821